CLINICAL TRIAL: NCT01502020
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Comparison Study to Determine the Therapeutic Equivalence of Generic Imiquimod Cream, 3.75% and Zyclara™ (Imiquimod) Cream, 3.75% in Subjects With Actinic Keratoses
Brief Title: A Bioequivalence Study With Clinical Endpoints Comparing Generic Imiquimod Cream, 3.75% and Zyclara™ (Imiquimod) Cream, 3.75% in Subjects With Actinic Keratoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actavis Mid-Atlantic LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 094-3152-301
Record Dates: First submitted 2011-12-23; First posted 2011-12-30 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Actinic Keratoses
Keywords: actinic keratoses; actinic keratosis; imiquimod, 3.75%; imiquimod; Zyclara; Actinic keratoses of the face or balding scalp
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zyclara™ (Active Comparator)
  Interventions: Drug: imiquimod cream, 3.75%
- Generic Imiquimod Cream, 3.75% (Experimental)
  Interventions: Drug: imiquimod cream, 3.75%
- Vehicle Cream (Placebo Comparator)
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: imiquimod cream, 3.75% — Dosage form: Topical Cream Dosage: 3.75% Frequency: The assigned test article was to be applied once daily for two 2-week treatment cycles separated by a 2-week no treatment interval Duration of Treatment: Two 2-week treatment cycles separated by a 2-week no-treatment period and an 8-week follow-up period.
  Arms: Zyclara™
Drug: Vehicle Cream — Dosage form: Topical Cream Dosage: Placebo Frequency: The assigned test article was to be applied once daily for two 2-week treatment cycles separated by a 2-week no treatment interval Duration of Treatment: Two 2-week treatment cycles separated by a 2-week no-treatment period and an 8-week follow-up period.
  Arms: Vehicle Cream
Drug: imiquimod cream, 3.75% — Dosage form: Topical Cream Dosage: 3.75% Frequency: The assigned test article was to be applied once daily for two 2-week treatment cycles separated by a 2-week no treatment interval Duration of Treatment: Two 2-week treatment cycles separated by a 2-week no-treatment period and an 8-week follow-up period.
  Arms: Generic Imiquimod Cream, 3.75%

SUMMARY:
Zyclara™ (imiquimod) Cream, 3.75% is approved by the FDA for the treatment of actinic keratoses on the full face or balding scalp. Zyclara is applied once daily for two, 2-week treatment cycles separated by a 2-week no treatment applied interval. A generic imiquimod cream, 3.75% has been developed by Actavis Mid-Atlantic LLC for the topical treatment of clinically typical, visible or palpable actinic keratoses (AK) of the full face or balding scalp.

The current clinical study is designed to evaluate the therapeutic equivalence of this formulation with the currently marketed Zyclara™ (imiquimod) cream, 3.75% formulation (Graceway Pharmaceuticals LLC).

ELIGIBILITY:
Inclusion Criteria:

* Subject was male or female, 18 years of age or older.
* Subject provided written informed consent.
* Subject was willing and able to apply the test article as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
* Subject had a clinical diagnosis of actinic keratoses (AK) with at least five (5) and no more than 20 clinically typical, visible or palpable AK lesions, each at least 4mm in diameter, in an area greater than 25cm2 on the face (excluding ears) or balding scalp, but not both.
* Subject was in good general health and free of any disease state or physical condition that might have impaired evaluation of AK lesions or which, in the investigator's opinion, exposed the subject to an unacceptable risk by study participation.
* If subject was a woman of childbearing potential (WOCBP), she must have had a negative urine pregnancy test (UPT) and agreed to use an effective form of birth control for the duration of the study (e.g., abstinence, stabilized on hormonal contraceptives for at least three months [oral, implant, injection, IUD, patch or NuvaRing] condom and spermicidal or diaphragm and spermicidal). Abstinence was an acceptable form of birth control for subjects who were not sexually active. Subjects who became sexually active during the trial had to agree to use an effective, non-prohibited form of birth control for the duration of the study.

Exclusion Criteria:

* Subject was pregnant, lactating, or planning to become pregnant during the study.
* Subjects had hyperkeratotic, hypertrophic or atypical AKs (e.g., AK > 1 cm2 in size) in the Treatment Area.
* Subject was enrolled in an investigational drug or device study during the study period.
* Subject was planning to be exposed to artificial tanning devices or excessive sunlight during the trial.
* Subject was immunosuppressed (e.g., HIV, systemic malignancy, graft vs. host disease, etc.).
* Subject had experienced an unsuccessful outcome from previous imiquimod therapy (An unsuccessful outcome was defined as after a reasonable therapeutic trial with no compliance issues, topical application did not work).
* Subject had used an investigational drug or investigational device within 30 days prior to the Baseline Visit.
* Subject had laser resurfacing, PUVA (Psoralen + ultraviolet A) therapy, UVB therapy, chemical peels or dermabrasion on the face or balding scalp within 6 months prior to the Baseline Visit.
* Subject had cryodestruction or chemodestruction, curettage, photodynamic therapy, surgical excision or other treatments for actinic keratosis on the face or scalp within one month prior to the Baseline Visit.
* Subject had used oral corticosteroid therapy, interferon, cytotoxic drugs, immunomodulators, immunosuppressive therapies or retinoids within one month prior to the Baseline Visit.
* Subject had used topical medications, corticosteroids, alpha hydroxy acids (e.g., glycolic acid, lactic acid etc. > 5%), beta hydroxy acid (salicylic acid > 2%), urea >5%, 5-fluorouracil, diclofenac, imiquimod or prescription retinoids (e.g., tazarotene, adapalene, tretinoin) to the face or balding scalp within one month prior to the Baseline Visit.
* Subject had used topical creams, lotions or gels of any kind to the selected Treatment Area within one day prior to the Baseline Visit.
* Subject had a basal cell or squamous cell carcinoma within the Treatment Area within one year of study enrollment.
* Subject had a history of sensitivity to any of the ingredients in the test articles.
* Subject had any skin pathology or condition (e.g., facial/scalp psoriasis, atopic dermatitis, acne, rosacea, etc.) that, in the investigator's opinion, could have interfered with the evaluation of the test article, worsened due to the treatment or required the use of interfering topical, systemic or surgical therapy.
* Subject had any condition which, in the investigator's opinion, would have made it unsafe or precluded the subject's ability to fully participate in the research study.
* Subject was known to be noncompliant or was unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Complete clearance rate | 8 weeks post treatment period
  Complete clearance rate (treatment success) was defined as the proportion of subjects in a treatment group with 100% clearance of all AK lesions within the Treatment Area. The primary efficacy endpoint was the proportion of subjects in the per-protocol (PP) population with treatment success at Week 14/EOS. All AKs (Baseline and new lesions), independent of size, within the Treatment Area were included in the AK lesion counts.
Dosing Compliance | 8 weeks post treatment period
  Measures of test article compliance included the total number of days of test article applications recorded on the CRFs and verified from the data in the subject diaries. Compliant subjects were defined as those who applied at least 75% and no more than 125% of the test article applications.
Adverse Events | 14 weeks
  The severity and frequency of adverse events (AEs) were assessed in the three treatment groups.
Local Skin Reactions | 14 weeks
  The severity and frequency of local skin reactions (LSRs) were assessed in the three treatment groups.

SECONDARY OUTCOMES:
Partial Clearance Rate | 8 weeks post treatment
  Partial clearance rate was defined as the proportion of subjects in a treatment group with 75% or more reduction in the AK count in the Treatment Area at Week 14/EOS as compared to Baseline.
Percent Change in the AK number | 8 weeks post treatment
  Percent change in the AK number as compared to Baseline at Week 14/EOS was a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Piacquadio, M.D., Study Director — Therapeutics, Inc.
Locations (19):
- United States (19):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - International Dermatology Research, Inc., Miami, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Indiana Clinical Trials Center, Plainfield, Indiana
  - Dermatology Specialists, Louisville, Kentucky
  - Michigan Center for Research Corp., Clinton Township, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, P.C., Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology, Laser & Vein Specialists of the Carolinas,, Charlotte, North Carolina
  - Dermatology Research Center of Cincinnati, Cincinnati, Ohio
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - DermResearch, Inc., Austin, Texas
  - Suzanne Bruce and Associates, P.A., Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas